CLINICAL TRIAL: NCT00321243
Title: Evaluation of a Four-Level Triage Scale (the Geneva Emergency Triage Scale) Using a Computer Triage Simulator
Brief Title: Evaluation of Emergency Triage Using a Computerized Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: O. Rutschmann, HUG, Geneva
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CER 05-213
Record Dates: First submitted 2006-02-06; First posted 2006-05-03 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Emergencies
Keywords: triage
MeSH Terms: conditions — Emergencies

INTERVENTIONS:
Behavioral: Visual clues

SUMMARY:
A four-level triage scale (the Geneva Emergency Triage Scale, GETS) has been used since 1997 in our emergency department (ED). A recent evaluation of this scale showed that our instrument had an excellent intra-rater reliability but insufficient inter-rater reliability. We also observed a wide variability in the way triage nurses perform (J Clin Epidemiology, 2006 in press). These variations in the triage process are mainly explained by a poor standardization of vital signs measurement. Therefore, we have recently modified our triage instrument and introduced explicit criteria for vital signs evaluation during the triage process.

The objectives of this study are:

* To evaluate the inter- and intra-rater reliability of our modified triage scale using a computer simulator
* To measure the impact of visual clues on the triage decisions when using the triage simulator
* To evaluate the performance of triage nurses and chief physicians in their triage decisions.

We expect to observe:

* an improvement of the inter-rater reliability of our instrument compared to the previous version
* a better standardization and more systematic use of vital signs measurement
* a higher reliability when visual clues are given to the evaluator
* lower rates of under- and over-estimation of emergency levels.

DETAILED DESCRIPTION:
A four-level triage scale (the Geneva Emergency Triage Scale, GETS) has been used since 1997 in our emergency department (ED). A recent evaluation of this scale showed that our instrument had an excellent intra-rater reliability but insufficient inter-rater reliability. We also observed a wide variability in the way triage nurses perform (J Clin Epidemiology, 2006 in press). These variations in the triage process are mainly explained by a poor standardization of vital signs measurement. Therefore, we have recently modified our triage instrument and introduced explicit criteria for vital signs evaluation during the triage process.

The objectives of this study are:

* To evaluate the inter- and intra-rater reliability of our modified triage scale using a computer simulator
* To measure the impact of visual clues on the triage decisions when using the triage simulator
* To evaluate the performance of triage nurses and chief physicians in their triage decisions.

We expect to observe:

* an improvement of the inter-rater reliability of our instrument compared to the previous version
* a better standardization and more systematic use of vital signs measurement
* a higher reliability when visual clues are given to the evaluator
* lower rates of under- and over-estimation of emergency levels.

ELIGIBILITY:
Inclusion Criteria:

* Triage nurses
* Emergency physicians

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Inter-rater and intra-rater reliability
Performance of evaluators

SECONDARY OUTCOMES:
Impact of visual clues on reliability

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland